CLINICAL TRIAL: NCT04287322
Title: Effect of Auditory and Tactile-kinesthetic Stimulation on Physiological Parameters, Physical Growth and Behaviour of Preterm Neonates
Brief Title: Effect of Auditory and Tactile-kinesthetic Stimulation on Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moi University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, CONSTANTINE OLIEBA AKWANALO, Clinical consultant, Moi University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOiU
Record Dates: First submitted 2020-02-18; First posted 2020-02-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Prematurity
Keywords: Maternal voice and tactile-kinesthetic stimulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Who Masked: Outcomes Assessor
Masking Description: The research assistants were blinded of aim of study, group allocations and interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tactile-kinesthetic stimulation (Experimental): Received tactile-kinesthetic stimulation three times a day (morning, afternoon and evening) for 10 days starting on day 3 of life (initial contact).
  Interventions: Behavioral: Tactile-kinesthetic stimulation
- Recorded maternal voice (Experimental): Listened to recorded maternal voice stimulation, three times a day (morning, afternoon and evening) for 10 days starting on day 3 of life (initial contact).
  Interventions: Behavioral: Recorded maternal voice
- Control (No Intervention): Received only standard nursery care

INTERVENTIONS:
Behavioral: Tactile-kinesthetic stimulation — Tactile-kinesthetic stimulation involved three sessions per day; morning, afternoon, and evening for 10 days starting day 3 of life (initial contact). The stimulation included three phases; Phase 1: With neonates in prone position, moderate pressure was used to provide 12 strokes with palms of the hands, each stroke lasting 5 seconds. The strokes were provided in each area as follows: head, neck, shoulders and back.
  Phase 2: In supine position, twelve moderate pressure strokes with palms of the hands, 5 seconds each, were provided in each area as follows:forehead,cheeks,chest, abdomen, upper limbs (each separately), lower limbs, palms and soles.
  Phase 3: Kinesthetic stimulation was done for 5 minutes. The intervention comprised five passive flexion and extension movements of each large joint.
  Arms: Tactile-kinesthetic stimulation
Behavioral: Recorded maternal voice — Following informed written consent from mothers,maternal voice was recorded (5 minutes talking to her baby and 10 minutes singing) using Philips Electronics, SA2RGA04KS, Netherlands. Recorded voice was played back inside the incubator or cot via micro audio system, which has been validated for safety and feasibility in previous studies (Doheny et al., 2012. Preterm neonate lay in supine/lateral position and recorded maternal voice was played for 15 minutes three times a day (morning, afternoon, evening) starting on day 3 of life up to day 12 of life (10 days).
  Arms: Recorded maternal voice

SUMMARY:
The study was conducted at a level II special care nursery of the Moi Teaching & Referral Hospital, an academic hospital in the Western region of Kenya. A sample of 108 preterm neonates who met eligibility criteria were studied (36 in auditory group, 36 in tactile-kinesthetic stimulation group, and 36 in control group). Auditory group listened to recorded maternal voice while tactile-kinesthetic group received massage and joint movements.The interventions were provided for 15 minutes, 3 times a day for 10 days while outcome measures were observed for 21 days. The neonates in the control group received standard neonatal care and were observed for outcome measures as those in the intervention groups.

DETAILED DESCRIPTION:
The study was aimed to determine the effect of auditory stimulation using recorded maternal voice and tactile-kinesthetic stimulation on physiological parameters, physical growth and behavioral development of preterm neonates. Three groups were involved; auditory stimulation, tactile-kinesthetic stimulation and control.

A quasi-experimental design was used to recruit 108 study subjects (36 in each group). A trained researcher conducted the stimulation in the intervention groups and two research assistants did the data entry. The research assistants were blinded to aim of study, group assignments, and interventions received by preterm neonates.

Preterm neonates baseline characteristics and clinical data were obtained at initial contact.

Physiological parameters (heart rate, oxygen saturation and body temperature) were monitored using a cardio-respiratory monitor (CODEC patient monitor CMS6000). Respiratory rate was measured by counting breaths per minute by the research assistant. The parameters were monitored and recorded before, during and after stimulation in the intervention groups. The control group had the measurement recorded in the morning, afternoon and evening.

Physical growth was assessed using weight measurement. Neonates are weighed daily in the nursery and data on weight was entered by research assistants on alternate days.

Neonatal behavioral assessment scale (NBAS) was used to assess behavior at initial contact, day 10, 17 and 24.

ELIGIBILITY:
Inclusion Criteria:

* on breast milk or formula feeds
* born 28 to 37 weeks gestational age
* ≥1000grams. The gestation was limited to ≥ 28 weeks and ≥1000grams based on significant neonatal mortality rate in neonates born before 28 weeks gestation and/or weighing <1000grams in MTRH (Njuguna et al., 2015).

Exclusion Criteria:

* critically ill and those on continuous positive airway pressure (CPAP)
* had neonatal infections including severe sepsis or necrotizing enterocolitis.

Ages: 3 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 15 minutes
  The preterm neonate was connected to a cardio-respiratory monitor (CODEC patient monitor CMS6000) and oxygen saturation readings were recorded by research assistant.
Heart rate | 15 minutes
  The preterm neonate was connected to a cardio-respiratory monitor (CODEC patient monitor CMS6000) and heart rate readings were recorded by research assistants.
Respiratory rate was measured by counting breaths per minute by the research assistants. | 15 minutes
  Recording respiratory rate
Body temperature | 15 minutes
  The preterm neonate was connected to a cardio-respiratory monitor (CODEC patient monitor CMS6000) with a temperature probe and temperature readings were recorded by research assistants.
Weight | 21 days
  Preterm neonates were weighed without clothes on ade digital weighing scale by the research assistants. The scale was disinfected, rechecked and caliberated to zero before each measurement.
Behavioral development | 21 days
  Neonatal Behavioral Assessment Scale by Brazelton TB & Nugent J., (2011) was administered to each preterm neonate in the study by a trained research assistant. Minimum score was 1 and maximum score 9, a higher score indicated better behavioral development of preterm neonate.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Esamai, PhD, Study Chair — Moi University
Locations (1):
- Constantine Akwanalo, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No